CLINICAL TRIAL: NCT02627313
Title: Tumor Bed Dose Delivery Using A Breast Specific Radiosurgery Device, The Gammapod: (A Clinical Feasibility Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTT-15-02
Record Dates: First submitted 2015-11-17; First posted 2015-12-10 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Breast Neoplasms
Keywords: Feasibility Studies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GammaPod (Experimental): GammaPod tumour bed boost
  Interventions: Device: GammaPod Tumour Bed Boost

INTERVENTIONS:
Device: GammaPod Tumour Bed Boost — Single fraction Tumour Bed boost of 8Gy in 1 Fraction

SUMMARY:
Conventional breast radiotherapy is delivered to the entirety of the breast in fractionated treatments given over several weeks. While these techniques are effective, there is a risk of late adverse events from irradiation of surrounding normal tissues and the protracted nature of the treatments is inconvenient to patients and resource-intensive for health care systems. There is an unmet need for novel treatments that can be delivered more quickly, with reduced normal tissue exposure, and without compromising efficacy. The GammaPod is a breast-specific radiotherapy delivery device that holds the promise in addressing these needs. Employing the engineering and physics principles from stereotactic radiotherapy, it allows delivery of a highly-localized radiation dose to a very limited volume of breast. The Ottawa Hospital is the only Canadian member of a consortium of five academic institutions that have acquired the GammaPod in order to rigorously evaluate its use in clinical trials. The aim of the current project is to complete a mandatory clinical feasibility study of the GammaPod as part of the application for Investigational Testing of Medical Devices from Health Canada. The study will focus on the use of the GammaPod to deliver a radiotherapy boost, that is, a localized dose of radiation just around the surgical bed, in a single treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must sign consent for study participation.
* The patient must be female and have a diagnosis of an invasive breast cancer that was treated surgically by a partial mastectomy.
* The surgical cavity is clearly visible on CT images and delineated by surgical clips
* We have at least one of the following clinico-pathological factors:

  * Age ≥18 and ≤ 50 years
  * Lymphovascular space invasion positive
  * Grade III histology
  * More than 2 close resection margins ( > 0 mm to ≤ 2 mm)
  * 1 close resection margin and extensive in-situ component (EIC)
  * Non-hormone sensitive breast cancer (ER and PR negative)
* Surgical margins are negative for invasive or non-invasive breast cancer.
* The volume of the TB PTV is less than 25% of the whole breast volume which is a criteria used for partial breast alone trials (NSABP B-39). The absolute value of the boost PTV is ≤ 100 cc
* Multifocal disease is allowed if it was removed by a single lumpectomy resection and the patient remained a candidate for breast conservation.
* Women of childbearing potential must use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills. For these women of childbearing potential, a negative pregnancy test must be obtained prior to study enrollment or waiver signed.
* The patient must weigh less than 150Kg (330lb), which is the limit of the imaging couch.
* The patient must be less than 6'6" in height.
* The patient must feel comfortable in the prone position.

Exclusion Criteria:

* Patients with proven multi-centric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm).
* Prior radiation therapy above the umbilicus
* Unable to fit into the immobilization breast cup with an adequate seal
* Male gender.
* Patient cannot comfortably be set up in the prone position (i.e. physical disability)
* Unable to fit into the breast immobilization device due to breast size or other anatomical reason.
* Mastectomy is the surgery performed.
* Patient has received prior radiotherapy to the involved breast.
* Regional nodal irradiation is part of the treatment plan.
* Tumor bed is less than 5 mm from the skin surface.
* Patients with skin involvement, regardless of tumor size.
* Patients with connective tissue disorders specifically systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Patients with psychiatric or addictive disorders as indicated in their medical histories that would preclude obtaining informed consent.
* Patients who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Treatment plan acceptability measured by the proportion of subjects with treatment plans deemed as acceptable, minor or major deviation. | Outcome measure on day 1 of radiation treatment
  Definition of treatment acceptability
  No deviation (acceptable): 100% prescription isodose surface covers at least 95% of the PTV. The near-minimum PTV dose (D98%) must be greater than 7.2 Gy and near-maximum PTV dose (D2%) must be less than 9.6 Gy.
  Minor deviation but acceptable: 95% prescription isodose surface covers between 95% and 100% of the PTV. No portion of the PTV receives <93% of the prescription dose. Near-maximum dose (D2%) to PTV exceeds prescription dose by >20% but <30%. All specified critical normal tissue DVH limits fall within 5% of the guidelines.
  Major deviations (unacceptable): 95% isodose surface covers < 95% of the PTV. A portion of PTV receives < 93% of the prescription dose. Near-maximum dose to PTV exceeds prescription dose by >30%. Any critical normal tissue DVH limit exceeds 5% of the specified value.